CLINICAL TRIAL: NCT06633874
Title: Smart Computing Models, Sensors, and Early Diagnostic Speech and Language Deficiencies Indicators in Child Communication
Acronym: SmartSpeech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Collaborators: DOTSOFT SA - GR (Unknown); TELEGLOBAL LP - GR (Unknown); Region of Epirus (Regional Operational Programme 'Epirus 2014-2020') - GR (Unknown); University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Eugenia I Toki, Associate Professor, SmartSpeech Scientific Project Manager, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HP1AB-28185 (MIS: 5033088); 18435/15.05.2020 (Registry Identifier: Research Ethics Committee, University of Ioannina)
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Developmental Language Disorders; Developmental Articulation Disorder; Speech Disorder; Neurodevelopmental Disorder (Diagnosis)
Keywords: screening; developmental speech and language disorders; speech disorder; language disorder; developmental disorder; developmental deficiencies; neurodevelopmental disorder; Early Diagnostic Speech and Language Deficiencies Indicators; Machine Learning; Neural Networks; Serious Game; Child Communication; neurodevelopmental screening
MeSH Terms: conditions — Language Development Disorders; Articulation Disorders; Speech Disorders; Neurodevelopmental Disorders; Disease; Language Disorders; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typically Developed Children PLAYING SERIOUS GAME (Experimental): The arm describes the data collection process to design an intelligent system that contributes to implementing new innovative tools to assist clinicians and/or other professionals in the complicated screening and diagnostic procedures for communication deficiencies in children.
  The main objective of this arm is to feed data from collected responses of TD children to the backend of the SmartSpeech system. The data we collect are Game responses, Speech responses, Gaze data from the tablet camera, and Heart Rate Variability (captured through the smartwatch). The backend system will use the data for training, evaluating, and validating the intelligence system.
  Interventions: Diagnostic Test: TD Playing the Serious Game APSOU
- Non-Typically Developed Children PLAYING SERIOUS GAME (Active Comparator): The arm describes the data collection process to design an intelligent system that contributes to implementing new innovative tools to assist clinicians and/or other professionals in the complicated screening and diagnostic procedures for communication deficiencies in children. The main objective of this arm is to feed data from collected responses of Non-TD children to the backend of the SmartSpeech system. The data we collect are Game responses, Speech responses, Gaze data from the tablet camera, and Heart Rate Variability (captured through the smartwatch). The backend system will use the data for training, evaluating, and validating the intelligence system.
  Interventions: Diagnostic Test: Non-TD Playing Serious Game

INTERVENTIONS:
Diagnostic Test: TD Playing the Serious Game APSOU — After parents participate in informative meetings, they proceed with written consent, SmartSpeech enrollment, and child developmental history. Then, the child may interact with the Serious Game. Typically developed (TD) children engage under the clinician's face-to-face supervision with the serious game APSOU, which assesses developmental domains, including speech, language, psychomotor, cognitive, psychoemotional, and hearing abilities. The average time for TD children to play the whole game is estimated to be 45 minutes.
  Arms: Typically Developed Children PLAYING SERIOUS GAME
Diagnostic Test: Non-TD Playing Serious Game — After parents participate in informative meetings, they proceed with written consent, SmartSpeech enrollment, and child developmental history. Then the child may interact with the serious game. Non-typically developed (non-TD) children engage under the clinician's face-to-face supervision with the serious game Apsou, which assesses developmental domains, including speech, language, psychomotor, cognitive, psychoemotional, and hearing abilities. The average time for non-TD children to play the whole game is estimated to be over an hour.
  Arms: Non-Typically Developed Children PLAYING SERIOUS GAME

SUMMARY:
This clinical trial aims to justify a protocol for designing and developing an automated decision-making system to support and enhance screening and early detection procedures for developmental speech/language difficulties in child communication. The system will utilize smart computing models, sensors, and early diagnostic speech and language deficiency indicators. The study participants will be typically and non-typically (neurodevelopmentally atypical) developing children, primarily in preschool and elementary school.

The key research questions the study seeks to address are:

1. Do differences exist between typically developing and neurodevelopmentally atypical children when engaging with the serious game used in the study?
2. If such differences are identified, can the collected data be utilized to train an automated decision-making system capable of accurately distinguishing between typically and neurodevelopmentally atypical children based on speech and language deficiencies?

Researchers will compare typically and non-typically developed children to see if the system can incorporate multiple data points from assessment domains to create a diagnostic profile.

After the parents are informed of the study and provide written consent, they enroll in the system. Participants will be asked to wear a smartwatch and play a serious game on a tablet under the supervision of a clinician. The system will collect data from the gameplay and sensors.

DETAILED DESCRIPTION:
In recent years, integrating digital and mobile technologies in health and education has opened new possibilities for monitoring and assessment. This study will build on these advancements by implementing artificial intelligence (AI) and machine learning models that offer real-time decision-making and personalized feedback. By automating critical aspects of the diagnostic process, this system will help bridge the gap between traditional clinical expertise and cutting-edge technology, ultimately enhancing early intervention efforts.

The SmartSpeech study will be a clinical trial designed to create and validate an automated decision-making system to enhance the screening and early detection of developmental speech and language difficulties in young children. This study will target typically and non-typically (neurodevelopmentally atypical) developing children, primarily focusing on preschool and elementary school-aged participants. The system will employ intelligent computing models, biometric sensors, and early diagnostic indicators of speech and language deficiencies to provide clinicians with a robust tool for identifying potential developmental issues.

Two primary research questions drive the trial:

1. Do differences exist between typically developing and neurodevelopmentally atypical children when engaging with the serious game used in the study?
2. If such differences are identified, can the collected data be utilized to train an automated decision-making system that accurately distinguishes between typically and neurodevelopmentally atypical children based on speech and language deficiencies?

To assess speech and language developmental skills and their manifestations, the interdisciplinary team will design a serious game (SG) based on theories that measure speech and language and psychomotor, cognitive, psychoemotional, and hearing skills. Each domain will assess the performance of specific tasks within the SG activities for the participant.

To address the questions of this study, data from typically developing children will be compared with data from non-typically developing children, analyzing whether the AI system can synthesize multiple data points across assessment domains to generate a comprehensive diagnostic profile.

Participants will be recruited through an open call distributed via private and public health and educational establishments across Greece. The recruitment process will focus on parents of typically and non-typically developing children aged 4 to 12. Parents will be invited to attend informational meetings where the objectives, procedures, and ethical guidelines of the study will be thoroughly explained.

During these sessions, parents will receive comprehensive information about the purpose of the study, including the specific role of the serious game developed in the study. The nature of the game, the expected involvement of their children, and the data collection methods will be discussed in detail to ensure transparency. Parents will be asked to provide informed written consent for their children to participate in full compliance with the General Data Protection Regulation and ethical considerations. These steps are essential to ensure that the rights and privacy of the participants will be protected throughout the study. Parents will also provide their child's developmental history in an online questionnaire embedded in the system.

The study will include typically developing preschool and school-aged children and non-typically developing children. It will not include children with other medical conditions or on medications that could potentially influence the results.

After an informative meeting and written consent from parents, participants will wear a smartwatch and engage in a serious game (designed and developed by the research team). Children will play the SG under the direct supervision of clinicians. This game will be designed to assess various developmental domains, including speech, language, psychomotor skills, cognitive function, psychoemotional behavior, and hearing abilities. The game will capture speech and language data through gameplay interactions alongside sensor data from the wearable device and the tablet camera (eye tracking and heart rate variability).

This game-based approach will naturally and engagingly collect diverse data points, ensuring a comprehensive evaluation of the child's speech and language abilities.

The system will form its datasets for analysis to detect speech and language development, feeding data into the selected artificial intelligence algorithms. The study will measure communication, psychomotor, cognitive, and psychoemotional skills through designed activities. The responses during gameplay will be evaluated, creating the developmental profile of the participant.

This structured and ethical recruitment process will ensure complete adherence to data protection and ethical standards while maintaining active engagement from both parents and children. By incorporating face-to-face supervision and real-time monitoring during gameplay, the study will guarantee the quality and integrity of the data collected for analysis.

The SG, paired with sensors from the smartwatch, will collect real-time data, including:

* Game responses
* Speech responses
* Gaze data from the tablet camera
* Heart Rate Variability (captured through the smartwatch)

This multi-modal data will be processed using neural network/machine learning algorithms to classify speech and language abilities across different developmental stages. The use of these advanced AI models will enable the system to:

* Identify patterns of speech/language deficiencies.
* Differentiate between typically and non-typically developed children.
* Create individualized diagnostic profiles for each participant.

Finally, an evaluation and verification of the intelligent system will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing preschoolers and school-aged children
* Children diagnosed with neurodevelopmental disorders
* Children should be native Greek speakers

Exclusion Criteria:

* Children with other medical conditions
* Children on medications that might affect the results of the study

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Speech and language for TD children | 10-20 minutes
  Score on Serious Game responses in Speech and language activities (0 - 100) by TD children
Psychomotor for TD children | 10-20 minutes
  Score on Serious Game responses in Psychomotor activities (0 - 100) by TD children
Cognitive for TD children | 10-20 minutes
  Score on Serious Game responses in Cognitive activities (0 - 100) by TD children
Psychoemotional for TD children | 10-20 minutes
  Score on Serious Game responses in Psychoemotional activities (0 - 100) by TD children
Hearing for TD children | 10-20 minutes
  Score on Serious Game responses in Hearing activities (0 - 100) by TD children
Eye-tracking fixation duration for TD children | 1-10 minutes
  Fixation Duration is the time the gaze stays on a single point in milliseconds (during specific activities in the Serious Game)
Eye-tracking trajectory path for TD children | 1-10 minutes
  Trajectory Path is the overall movement path of the gaze in millimeters on screen (during specific activities in the Serious Game)
Heart rate variability for TD children | 1-10 minutes
  Heart rate variability during the game that is calculated by HRV=(HRe-HRs)/HRs, HRs: Heart Rate at the start of the measurement, HRe: Heart Rate at the end of the measurement. The duration between start - end of each activity measurement is a few seconds
Speech and language for non-TD children | 10-20 minutes
  Score on Serious Game responses in Speech and language activities (0 - 100) by non-TD children
Psychomotor for non-TD children | 10-20 minutes
  Score on Serious Game responses in Psychomotor activities (0 - 100) by non-TD children
Cognitive for non-TD children | 10-20 minutes
  Score on Serious Game responses in Cognitive activities (0 - 100) by non-TD children
Psychoemotional for non-TD children | 10-20 minutes
  Score on Serious Game responses in Psychoemotional activities (0 - 100) by non-TD children
Hearing for non-TD children | 10-20 minutes
  Score on Serious Game responses in Hearing activities (0 - 100) by non-TD children
Eye-tracking fixation duration for non-TD children | 1-10 minutes
  Fixation Duration is the time the gaze stays on a single point in milliseconds (during specific activities in the Serious Game)
Eye-tracking trajectory path for non-TD children | 1-10 minutes
  Trajectory Path is the overall movement path of the gaze in millimeters on screen (during specific activities in the Serious Game)
Heart rate variability for non-TD children | 1-10 minutes
  Heart rate variability during the game that is calculated by HRV=(HRe-HRs)/HRs, HRs: Heart Rate at the start of the measurement, HRe: Heart Rate at the end of the measurement. The duration between start - end of each activity measurement is a few seconds

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia I Toki, PhD, Study Chair — University of Ioannina, Greece
Locations (1):
- University of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No
The participants of this study did not give written consent for their data to be shared publicly, so due to privacy restrictions and the sensitive nature of this research data sharing is not applicable

REFERENCES:
- [Derived] Toki EI, Zakopoulou V, Tatsis G, Pange J. Automated Detection of Neurodevelopmental Disorders Using Face-to-Face Mobile Technology Among Typically Developing Greek Children: Randomized Controlled Trial. JMIR Form Res. 2024 Oct 11;8:e53465. doi: 10.2196/53465. PMID 39393054